CLINICAL TRIAL: NCT01118091
Title: Prospective Randomized Comparative Study of Cell Transfer Therapy Using Short-Term Cultured Anti-Tumor Autologous Lymphocytes Following a Non-Myeloablative Lymphocyte Depleting Chemotherapy Regimen Compared to High-dose Aldesleukin in Metastatic Melanoma
Brief Title: Prospective Randomized Comparative Study of Cell Transfer Therapy Using CD8+-Enriched Short-Term Cultured Anti-Tumor Autologous Lymphocytes Following a Non-Myeloablative Lymphocyte Depleting Chemotherapy Regimen Compared to High-Dose Aldesleukin in M...
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 100117; 10-C-0117
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Skin Cancer; Melanoma; Metastatic Melanoma
Keywords: Immunotherapy; Metastatic Melanoma; Randomized; Cell Therapy; Skin Cancer; Melanoma
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1-Aldesleukin (Active Comparator): Aldesleukin 720,000 IU/kg IV over 15 minute every eight hours and continuing for up to 5 days (maximum of 15 doses). Patients will receive one additional cycle of aldesleukin approximately 10-14 days after completion of the first cycle of aldesleukin.
  Interventions: Biological: Aldesleukin
- Arm 2 - Adoptive cell therapy (Experimental): Adoptive Cell Therapy consisting of the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide, followed by infusion of between 1x10^9 to 2x10^11 CD8+ enriched tumor infiltrating lymphocytes (minimum of 5 x10^8) and the administration of high-dose aldesleukin.
  Interventions: Biological: CD8 enriched Young TIL

INTERVENTIONS:
Biological: Aldesleukin — Aldesleukin 720,000 IU/kg IV over 15 minute every eight hours and continuing for up to 5 days (maximum of 15 doses). Patients will receive one additional cycle of aldesleukin approximately 10-14 days after completion of the first cycle of aldesleukin.
  Arms: Arm 1-Aldesleukin
Biological: CD8 enriched Young TIL — Adoptive Cell Therapy consisting of the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide, followed by infusion of between 1x10^9 to 2x10^11 CD8+ enriched tumor infiltrating lymphocytes (minimum of 5 x 10^8) and the administration of high-dose aldesleukin.
  Arms: Arm 2 - Adoptive cell therapy

SUMMARY:
Background:

- Adoptive cell therapy involves taking white blood cells called lymphocytes from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient to allow the cells to attack the tumor. Because this process is lengthy and difficult to perform, researchers have been developing improved means of performing adoptive cell therapy. Researchers are now interested in comparing adoptive cell therapy with the standard treatment for metastatic melanoma (skin cancer).

Objectives:

- To compare the effectiveness of adoptive cell therapy with standard high-dose aldesleukin as a treatment for metastatic melanoma.

Eligibility:

* Individuals 18 years of age or older who have been diagnosed with metastatic melanoma and have not previously received aldesleukin therapy or cell therapy for their disease.
* Participants must have at least one tumor that can be easily removed as part of the treatment procedure.

Design:

* Participants will be screened with a full medical history, physical examination, blood and urine tests, and imaging scans to evaluate tumor size and treatment options.
* Participants will be separated into two groups, in which one group will have adoptive cell therapy and one will have aldesleukin treatment.
* Adoptive Cell Therapy

  * Participants will have a tumor sample taken in order to collect white blood cells for treatment. Participants whose tumors do not provide sufficient white blood cells may be switched to the aldesleukin-only treatment group.
  * The white blood cells will be grown in the laboratory for several weeks.
  * Prior to receiving cell therapy, participants will receive chemotherapy for 7 days to improve the chances of successful treatment.
  * Participants will have cell therapy followed by high-dose aldesleukin treatment every 8 hours for up to 5 days. This treatment will be followed by 1 to 2 weeks of recovery time as an inpatient at the clinical center.
  * Participants will be evaluated at 12 weeks following the start of the study, every 2 to 3 months for the first year, every 6 months for the next 5years, and then yearly thereafter..
* Standard Aldesleukin Treatment

  * Participants will have high-dose aldesleukin treatment every 8 hours for up to 5 days (one cycle of treatment), and will have a second cycle of treatment 7 to 10 days after the first cycle.
  * If tests show that the tumors have grown, participants will be offered the chance to have additional cycles of aldesleukin, or begin a cell therapy treatment.
* Participants will be evaluated at 12 weeks following the start of the study, every 2 to 3 months for the first year, every 6 months for the next 5years, and then yearly thereafter.

DETAILED DESCRIPTION:
Background:

* Tumor Infiltrating Lymphocytes (TIL) can mediate the regression of bulky metastatic melanoma when administered to the autologous patient along with high-dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting chemotherapy preparative regimen.
* Although this adoptive cell therapy (ACT) has been shown capable of mediating objective clinical responses in patients with metastatic melanoma, including patients who have previously been treated with aldesleukin or chemotherapy, the treatment is only available in the Surgery Branch, National Cancer Institute (NCI) and in just one or two other institutions in the United States.
* Despite our reports of the objective regressions in patients receiving adoptive cell therapy (ACT), doubts have been raised concerning the possible influence of patient selection bias that may have accounted for the increase in survival using ACT compared to historical controls.
* ACT is a cumbersome and labor intensive procedure which has discouraged many from applying it. We have recently developed simplifications in the technique for generating TIL that are also capable of mediating objective responses.
* To evaluate the efficacy of ACT we are now proposing a prospective randomized trial to compare this form of therapy with standard available treatment for patients with metastatic melanoma.

Objectives:

* To determine, in a prospective randomized trial, the response rate and progression free survival of patients with metastatic melanoma receiving either ACT or standard high-dose aldesleukin treatment.
* Survival rate will be evaluated as a secondary endpoint.
* To determine the toxicity of these two treatment regimens.

Eligibility:

Patients who are 18 years of age or older must have:

* Evaluable metastatic melanoma;
* No prior treatment with high-dose aldesleukin (greater than or equal to 600,000 IU IL-2 q8h or the equivalent)
* No contraindications to high-dose aldesleukin administration;
* No concurrent major medical illnesses or any form of immunodeficiency;
* Lesions of at least 2cm in diameter that can be surgically removed with minimal morbidity.

Design:

* Prior to amendment D, patients with metastatic melanoma lesions that can be resected with minimal morbidity will be prospectively randomized to receive either ACT using CD8+ young TIL (arm 2) and aldesleukin (arm 1) following a non-myeloablative chemotherapy preparative regimen, or will receive standard high-dose aldesleukin therapy.
* With the approval of amendment D, arm 1 and 2 will be closed, and two new arms will be opened. Patients with metastatic melanoma lesions that can be resected with minimal morbidity will be prospectively randomized to receive either ACT using young TIL (arm 4) and aldesleukin (arm 3) following a non-myeloablative chemotherapy preparative regimen, or will receive standard high-dose aldesleukin therapy.
* Response rate and time to progression will be evaluated for all patients on an intent-to-treat basis.
* Patients may crossover to the other treatment arm after progressive disease is documented by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, if still eligible.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic melanoma with at least one lesion that is resectable for tumor infiltrating lymphocytes (TIL) generation. The lesion must be of at least 2cm in diameter that can be surgically removed with minimal morbidity (defined as any operation for which expected hospitalization is less than or equal to 7 days).
  2. Patients with 3 or less brain metastases are eligible. Note: If lesions are symptomatic or greater than or equal to 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible.
  3. No prior high-dose aldesleukin therapy at a dose of greater than or equal to 600,000 IU/kg.
  4. Greater than or equal to 18 years of age.
  5. Willing to practice birth control during treatment and for four months after receiving all protocol related therapy.
  6. Life expectancy of greater than three months.
  7. Willing to sign a durable power of attorney.
  8. Able to understand and sign the Informed Consent Document.
  9. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  10. Hematology:
* Absolute neutrophil count greater than 1000/mm^3 without support of filgrastim
* Normal White blood cell (WBC) (> 3000/mm^3).
* Hemoglobin greater than 8.0 g/dl
* Platelet count greater than 100,000/mm^3

  k. Serology:
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, or hepatitis C antibody or antigen.

  l. Chemistry:
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than three times the upper limit of normal.
* Calculated creatinine clearance estimated glomerular filtration rate(eGFR) > 50 ml/min.
* Total bilirubin less than or equal to 2 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dl.

  m. More than four weeks must have elapsed since any prior systemic therapy at the time the time of randomization, and patients' toxicities must have recovered to a grade 1 or less (except for alopecia or vitiligo). Patients must have stable or progressing disease after prior treatment. Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria.

  n. Six weeks must have elapsed since any prior anti-CTLA4 antibody therapy to allow antibody levels to decline.

  o. Patients who have previously received any cytotoxic T-lymphocyte antigen 4 (anti-CTLA4) antibody and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Prior cell transfer therapy which included a non-myeloablative or myeloablative chemotherapy regimen.
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Systemic steroid therapy requirement.
4. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
5. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and Acquired Immunodeficiency Syndrome (AIDS)).
6. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization or ischemic symptoms.
9. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
10. In patients > 60 years old, documented LVEF of less than or equal to 45%.
11. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking
    * Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaprasad Srinivasan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Atkins MB, Kunkel L, Sznol M, Rosenberg SA. High-dose recombinant interleukin-2 therapy in patients with metastatic melanoma: long-term survival update. Cancer J Sci Am. 2000 Feb;6 Suppl 1:S11-4. PMID 10685652
- [Background] Kirkwood MW, Yeates KO, Taylor HG, Randolph C, McCrea M, Anderson VA. Management of pediatric mild traumatic brain injury: a neuropsychological review from injury through recovery. Clin Neuropsychol. 2008 Sep;22(5):769-800. doi: 10.1080/13854040701543700. Epub 2007 Sep 1. PMID 17896204

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Aldesleukin: Aldesleukin 720,000 IU/kg IV over 15 minute every eight hours and continuing for up to 5 days (maximum of 15 doses). Patients will receive one additional cycle of aldesleukin approximately 10-14 days after completion of the first cycle of aldesleukin.
  Aldesleukin : Aldesleukin 720,000 IU/kg IV over 15 minute every eight hours and continuing for up to 5 days (maximum of 15 doses). Patients will receive one additional cycle of aldesleukin approximately 10-14 days after completion of the first cycle of aldesleukin.
- Arm 2 - Adoptive Cell Therapy: Adoptive Cell Therapy consisting of the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide, followed by infusion of between 1x10^9 to 2x10^11 CD8+ enriched tumor infiltrating lymphocytes (minimum of 5 x10^8) and the administration of high-dose aldesleukin.
  CD8 enriched Young TIL : Adoptive Cell Therapy consisting of the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide, followed by infusion of between 1x10^9 to 2x10^11 CD8+ enriched tumor infiltrating lymphocytes (minimum of 5 x 10^8) and the administration of high-dose aldesleukin.
Period: Overall Study
Arm/Group | Arm 1 - Aldesleukin | Arm 2 - Adoptive Cell Therapy
Started | 7 (2pts were randomized to Arm 2, were not able to grow cell product, were treated with Arm 1 regimen.) | 5
Completed | 7 (Continued from above: These 2 pts are only represented in Arm 1 (and not Arm 2).) | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Aldesleukin | Arm 2 - Adoptive Cell Therapy | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (8.2) | 53.6 (9.5) | 49.15 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response (CR) is the disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 3 years
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Aldesleukin | Arm 2 - Adoptive Cell Therapy
Number analyzed (Participants) | 7 | 5
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 1
  Progressive Disease | 6 | 4
  Stable Disease | 0 | 0

2. Secondary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 3 years
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Aldesleukin | Arm 2 - Adoptive Cell Therapy
Number analyzed (Participants) | 7 | 5
Participants | 7 | 5

3. Primary Outcome: Progression Free Survival
Description: Measured from the time of randomization to time of progression (or death).
Time Frame: 3 years
Measure: Number; unit: Days
Arm/Group | Arm 1 - Aldesleukin | Arm 2 - Adoptive Cell Therapy
Number analyzed (Participants) | 7 | 5
Days
  Patient 1 | 307 | 0
  Patient 2 | 0 | 130
  Patient 3 | 0 | 88
  Patient 4 | 0 | 174
  Patient 5 | 54 | 0
  Patient 6 | 0 | 88
  Patient 7 | 129 | 0
  Patient 8 | 0 | 515
  Patient 9 | 117 | 0
  Patient 10 | 279 | 0
  Patient 11 | 58 | 0
  Patient 12 | 130 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 - Aldesleukin | Arm 2 - Adoptive Cell Therapy
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Aldesleukin (N=7) | Arm 2 - Adoptive Cell Therapy (N=5)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 6 (7) | 5 (7)
Hypotension (Cardiac disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Acute vascular leak syndrome (Vascular disorders) | 1 (1) | 2 (3)
Platelets (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Pain (General disorders) | 3 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Cardiac arrhythmia - Other, Specify, (Cardiac disorders) | 1 (1) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (2) | 0 (0)
Neuropathy-sensory (Nervous system disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Neutrophilis/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Febrile neutropenia (fever of unknown origin with (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No